CLINICAL TRIAL: NCT07300072
Title: Pneumothorax Risk and Pleural-Depth-Trimmed Hookwire: A Retrospective Cohort Study With Propensity Score Matching in Preoperative CT-Guided Lung Nodule Localization
Brief Title: Pneumothorax Safety of Pleural-Depth-Trimmed Hookwires for Lung Nodule Localization
Status: Completed | Type: Observational
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Guo-Zhi Wang, Attending Physician, Chung Shan Medical University
Other Study IDs: CS2-25160
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Nodules; Pneumothorax Iatrogenic Postprocedural; Propensity Score Matching
Keywords: Pneumothorax; Lung nodule localization; Pleural-Depth-Trimmed Hookwire; Propensity score matching
MeSH Terms: conditions — Pneumothorax | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Hookwire-Localized: This group consists of lung nodules that were localized using the Pleural-Depth-Trimmed Hookwire (Hawkins II breast localization needles, pre-trimmed to exceed the nodule-to-pleura depth by 5 mm to10 mm) combined with dye tattoos. This approach was primarily used for target lesions located >30 mm from the pleura. In the PSM analysis, this group served as the intervention group (n=237).
  Interventions: Procedure: Preoperative CT-Guided Lung Nodule Localization with Pleural-Depth-Trimmed Hookwire (PDTH) Technique
- Non-Hookwire-Localized: This group consists of lung nodules localized using only the Patent Blue Vital Dye. This method was used for target lesions located within 20 mm of the pleura. In the PSM analysis, this group served as the comparison group (n=237).
  Interventions: Procedure: Preoperative CTGuided Lung Nodule Localization with Patent Blue Vital Dye (PBVD) Localization Technique

INTERVENTIONS:
Procedure: Preoperative CT-Guided Lung Nodule Localization with Pleural-Depth-Trimmed Hookwire (PDTH) Technique — The PDTH Technique is a modified localization method using the U.S. FDA-regulated Hawkins II hookwire (Argon Medical Devices, US).
  The standard wire is pre-trimmed to only exceed the nodule-to-pleura depth by a minimal 5 mm to 10 mm. This crucial modification aims to reduce iatrogenic pneumothorax risk by preventing excessive wire length from protruding and causing pleural friction or trauma during the procedure.
  This technique is primarily used for deeper lesions (>30 mm from the pleura) and is integrated with the Laser Angle Guide Assembly (LAGA) system to ensure precise needle insertion and a dual patent blue vital dye tattooing strategy.
  Groups: Hookwire-Localized
Procedure: Preoperative CTGuided Lung Nodule Localization with Patent Blue Vital Dye (PBVD) Localization Technique — This intervention serves as the comparison group for the Pleural-Depth-Trimmed Hookwire (PDTH) technique in the Propensity Score Matching (PSM) analysis. This localization method utilizes only a vital dye marker and is generally associated with a lower complication risk due to its non-solid nature.
  Localization Marker: Patent blue vital dye (PBVD; Guerbet, France, 2.5%).
  Indication: The dye-only method was typically used for target lesions located within 20 mm of the pleura.
  Procedure: Two dye tattoos were marked on the lung parenchyma using a thinner 23-gauge, 89 mm spinal needle or a 23-gauge, 70 mm spinal needle.
  Guidance: Procedures were conducted under CT guidance, utilizing the Laser Angle Guide Assembly (LAGA) system.
  Purpose: In the context of this study, this group provides the benchmark comparison to determine the non-inferiority of the PDTH technique regarding the risk of iatrogenic pneumothorax.
  Groups: Non-Hookwire-Localized

SUMMARY:
The goal of this observational study is to learn about the pneumothorax risk associated with the Pleural-Depth-Trimmed Hookwire (PDTH) technique in patients undergoing Preoperative CT-Guided Lung Nodule Localization (POCTGL). The main question it aims to answer is: Does the specialized PDTH technique increase the risk of iatrogenic pneumothorax compared to dye-only localization in a setting utilizing advanced puncture guidance?. Participants were a retrospective cohort of patients who underwent POCTGL procedures between 2015 and 2022, and their procedural data and post-procedural complications were analyzed.

DETAILED DESCRIPTION:
The unique contribution of this retrospective cohort study lies in its rigorous evaluation of an institutional, multi-component protocol for Preoperative CT-Guided Lung Nodule Localization (POCTGL), specifically focusing on the safety of the Pleural-Depth-Trimmed Hookwire (PDTH) technique when used in conjunction with the Laser Angle Guide Assembly (LAGA) system.

Specialized Intervention Technique Pleural-Depth-Trimmed Hookwire (PDTH)

Technical Rationale: The PDTH technique was developed to mitigate the high pneumothorax risk (historically reported up to 35%) associated with standard hookwires. This risk is hypothesized to result from the excessive length of the traditional hookwire protruding from the chest wall, causing friction and pleural trauma during patient movement and respiration.

Execution: The standard localization hookwire (Hawkins II) is pre-trimmed prior to insertion. Its length is adjusted to only exceed the measured distance from the pleural surface to the target nodule by a minimal margin (5 mm∼10 mm), effectively eliminating the long, protruding segment.

Combined Approach: For deep lesions (typically >30 mm from the pleura), the PDTH is used in combination with a dual patent blue vital dye (PBV) tattooing strategy, providing multiple locational markers for the subsequent Video-Assisted Thoracoscopic Surgery (VATS).

Laser Angle Guide Assembly (LAGA)

The protocol incorporates the LAGA system, a device that provides visual, objective guidance for the needle trajectory. This system's primary benefit is to improve the accuracy of the initial puncture, which directly correlates with reducing the number of puncture attempts, a critical modifiable risk factor for pneumothorax confirmed by this study.

Rigorous Statistical Methodology

To provide a robust comparison despite the non-randomized, observational nature of the data, the study employed advanced statistical methods:

Generalized Estimating Equations (GEE): Used to identify independent risk factors for pneumothorax across the entire cohort. GEE was crucial for accounting for the non-independence of observations, as many patients underwent multiple procedures or had multiple nodules localized within a single session.

Propensity Score Matching (PSM): Utilized to control for selection bias inherent in marker choice (PDTH vs. dye-only). PSM was performed strictly on the first-localized nodule from each procedure, employing a 1:1 nearest-neighbor match, adjusted for key confounding variables like lobe location and specific patient position.

Clinical Implications

The study reports an overall iatrogenic pneumothorax rate of 5.6%, which is substantially lower than historical data, supporting the efficacy of the comprehensive protocol. Crucially, both GEE and PSM analyses confirmed that the use of the PDTH technique was not associated with an increased risk of pneumothorax compared to the dye-only localization group (PSM comparison: p=0.662), validating the specialized, modified hookwire technique as a safe option within this low-risk protocol.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive series of patients who underwent Preoperative Computed Tomography-Guided Lung Nodule Localization (POCTGL) at our medical center between September 2015 and January 2022.
* All included procedures were performed in patients who subsequently underwent Video-Assisted Thoracoscopic Surgery (VATS) lung resection on the same day.

Exclusion Criteria For the primary Generalized Estimating Equations (GEE) analysis:

* Nodules localized after a pneumothorax event occurred (n=59) were excluded.

Exclusion Criteria For the Propensity Score Matching (PSM) analysis:

* Nodules localized after a pneumothorax event (n=59).
* Nodules that were not the first localized nodule during the POCTGL procedure (n=495).
* Nodules associated with a previous ipsilateral VATS (n=16).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The final analysis cohort included 1,072 POCTGL procedures. The procedures resulted in 1,567 evaluable lung nodules after the initial exclusion.
  Demographics: The median age was 55 years (IQR, 48-63). The cohort was predominantly women (74.6%) and nonsmokers (86.3%).
  Lesion Characteristics: The median lesion size was 6.5 mm (IQR, 5.0-8.0) , with a median depth from the pleura of 19 mm (IQR, 10.0-30.0).
  Procedure Type: Most procedures (90.3%) were for initial VATS , and the majority involved a single lesion (65.5%).
Sampling Method: Non-Probability Sample
Enrollment: 1072 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Iatrogenic Pneumothorax Rate | Immediately following the localization procedure, documented on the final confirmatory CT scan.
  The primary outcome is the incidence of iatrogenic pneumothorax documented as air presence on post-localization Computed Tomography (CT) scans. Pneumothorax was considered significant if the airspace thickness exceeded 3 cm. The rate was assessed to identify independent risk factors and to compare the safety of the Pleural-Depth-Trimmed Hookwire (PDTH) technique against non-hookwire localization.

SECONDARY OUTCOMES:
Requirement for Catheter Aspiration | Immediately post-localization, during the POCTGL procedure documentation.
  The rate of procedures requiring therapeutic intervention (catheter aspiration) for severe pneumothorax, defined as an airspace thickness exceeding 3 cm.
Incidence of Other Adverse Events | Documented in real-time during the POCTGL procedure.
  The incidence rate of other documented complications at the time of the POCTGL procedures. These complications included intolerable pain, severe cough, dizziness, and hookwire dislodgement.
Technical Factors Associated with Pneumothorax | Assessed based on real-time procedural data collected during the POCTGL procedure.
  Identifying independent risk factors (e.g., number of puncture attempts, lesion order, patient position) associated with increased odds of pneumothorax using Generalized Estimating Equations (GEE) .

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) are not publicly available due to patient confidentiality and ethical restrictions. However, de-identified IPD supporting the findings of this study will be made available upon request. Researchers who meet the criteria for access to confidential data may submit requests to the Institutional Review Board (IRB) of Chung Shan Medical University Hospital, Taichung, Taiwan, for review and approval.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Start Date: Upon request, 90 days after publication. End Date: Five years following study publication.
Access Criteria: Access to the de-identified Individual Participant Data (IPD) and supporting documentation (e.g., Statistical Analysis Plan and Analytic Code ) will be considered for qualified researchers who meet the criteria for accessing confidential data.
  Who: Qualified researchers who submit a detailed research proposal and sign a data access agreement.
  What: De-identified IPD supporting the findings, along with the study protocol and statistical analytic code.
  How: Requests must be submitted to the Institutional Review Board (IRB) of Chung Shan Medical University Hospital, Taichung, Taiwan, for formal review and approval. Access will be granted following a privacy risk assessment by the IRB and/or relevant institutional committees.
URL: https://web.csh.org.tw/web/221000/?page_id=5073

REFERENCES:
- [Background] Huang JY, Tsai SC, Wu TC, Lin FC. Puncture frequency predicts pneumothorax in preoperative computed tomography-guided lung nodule localization for video-assisted thoracoscopic surgery. Thorac Cancer. 2022 Jul;13(13):1925-1932. doi: 10.1111/1759-7714.14457. Epub 2022 May 25. PMID 35614380
- [Background] Tsai SC, Wu TC, Lai YL, Lin FC. Preoperative computed tomography-guided pulmonary nodule localization augmented by laser angle guide assembly. J Thorac Dis. 2019 Nov;11(11):4682-4692. doi: 10.21037/jtd.2019.10.60. PMID 31903257
- [Background] Lin FC, Tsai SC, Tu HT, Lai YL, Wu TC. Computed tomography-guided localization with laser angle guide for thoracic procedures. J Thorac Dis. 2018 Jun;10(6):3824-3828. doi: 10.21037/jtd.2018.05.162. PMID 30069383
- [Background] Wang J, Yao J, Xu L, Shan L, Zhai R, Gao L, Liu L, Yao F. Comparison of cyanoacrylate and hookwire for localizing small pulmonary nodules: A propensity-matched cohort study. Int J Surg. 2019 Nov;71:49-55. doi: 10.1016/j.ijsu.2019.09.001. Epub 2019 Sep 12. PMID 31521836
- [Background] Sun X, Fu J, Ma C, Song Z, Yang S, Jin L, Duan F. CT-guided microcoil versus hook-wire localization of pulmonary nodule prior to video-assisted thoracoscopic surgery without fluoroscopic guidance. BMC Pulm Med. 2024 Oct 8;24(1):492. doi: 10.1186/s12890-024-03306-0. PMID 39379924
- [Background] Han R, Wang LF, Teng F, Lin J, Xian YT, Lu Y, Wu AL. Presurgical computed tomography-guided localization of lung ground glass nodules: comparing hook-wire and indocyanine green. World J Surg Oncol. 2024 Feb 10;22(1):51. doi: 10.1186/s12957-024-03331-7. PMID 38336734
- [Background] Chu S, Wei N, Lu D, Chai J, Liu S, Lv W. Comparative study of the effect of preoperative hookwire and methylene blue localization techniques on post-operative hospital stay and complications in thoracoscopic pulmonary nodule surgery. BMC Pulm Med. 2022 Sep 5;22(1):336. doi: 10.1186/s12890-022-02129-1. PMID 36064381
- [Background] Yang F, Zhao H, Sui X, Zhang X, Sun Z, Zhao X, Wang J. Comparative study on preoperative localization techniques using microcoil and hookwire by propensity score matching. Thorac Cancer. 2020 Jun;11(6):1386-1395. doi: 10.1111/1759-7714.13365. Epub 2020 Mar 24. PMID 32207226
- [Background] Yamagami T, Terayama K, Yoshimatsu R, Matsumoto T, Miura H, Nishimura T. Role of manual aspiration in treating pneumothorax after computed tomography-guided lung biopsy. Acta Radiol. 2009 Dec;50(10):1126-33. doi: 10.3109/02841850903232707. PMID 19922309
- [Background] Park CH, Han K, Hur J, Lee SM, Lee JW, Hwang SH, Seo JS, Lee KH, Kwon W, Kim TH, Choi BW. Comparative Effectiveness and Safety of Preoperative Lung Localization for Pulmonary Nodules: A Systematic Review and Meta-analysis. Chest. 2017 Feb;151(2):316-328. doi: 10.1016/j.chest.2016.09.017. Epub 2016 Oct 4. PMID 27717643
- [Background] Zaman M, Bilal H, Woo CY, Tang A. In patients undergoing video-assisted thoracoscopic surgery excision, what is the best way to locate a subcentimetre solitary pulmonary nodule in order to achieve successful excision? Interact Cardiovasc Thorac Surg. 2012 Aug;15(2):266-72. doi: 10.1093/icvts/ivs068. Epub 2012 May 9. PMID 22572410
- [Background] Nakashima S, Watanabe A, Obama T, Yamada G, Takahashi H, Higami T. Need for preoperative computed tomography-guided localization in video-assisted thoracoscopic surgery pulmonary resections of metastatic pulmonary nodules. Ann Thorac Surg. 2010 Jan;89(1):212-8. doi: 10.1016/j.athoracsur.2009.09.075. PMID 20103238
- [Background] Saito H, Minamiya Y, Matsuzaki I, Tozawa K, Taguchi K, Nakagawa T, Hashimoto M, Hirano Y, Ogawa J. Indication for preoperative localization of small peripheral pulmonary nodules in thoracoscopic surgery. J Thorac Cardiovasc Surg. 2002 Dec;124(6):1198-202. doi: 10.1067/mtc.2002.127331. PMID 12447187
- [Background] Suzuki K, Nagai K, Yoshida J, Ohmatsu H, Takahashi K, Nishimura M, Nishiwaki Y. Video-assisted thoracoscopic surgery for small indeterminate pulmonary nodules: indications for preoperative marking. Chest. 1999 Feb;115(2):563-8. doi: 10.1378/chest.115.2.563. PMID 10027460
- [Background] Chang GC, Chiu CH, Yu CJ, Chang YC, Chang YH, Hsu KH, Wu YC, Chen CY, Hsu HH, Wu MT, Yang CT, Chong IW, Lin YC, Hsia TC, Lin MC, Su WC, Lin CB, Lee KY, Wei YF, Lan GY, Chan WP, Wang KL, Wu MH, Tsai HH, Chian CF, Lai RS, Shih JY, Wang CL, Hsu JS, Chen KC, Chen CK, Hsia JY, Peng CK, Tang EK, Hsu CL, Chou TY, Shen WC, Tsai YH, Tsai CM, Chen YM, Lee YC, Chen HY, Yu SL, Chen CJ, Wan YL, Hsiung CA, Yang PC; TALENT Investigators. Low-dose CT screening among never-smokers with or without a family history of lung cancer in Taiwan: a prospective cohort study. Lancet Respir Med. 2024 Feb;12(2):141-152. doi: 10.1016/S2213-2600(23)00338-7. Epub 2023 Nov 29. PMID 38042167
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641